CLINICAL TRIAL: NCT04098887
Title: A Phase I Trial of Lattice Stereotactic Body Radiation Therapy (Lattice SBRT) for Localized Unresectable or Metastatic Conventional Type Chondrosarcoma
Brief Title: Lattice Stereotactic Body Radiation Therapy (Lattice SBRT) for Localized Unresectable or Metastatic Conventional Type Chondrosarcoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator decided to not go forward with the study.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-x296
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Chondrosarcoma
MeSH Terms: conditions — Chondrosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lattice stereotactic body radiation therapy (Experimental): Patients with up to 10 chondrosarcoma lesions will undergo radiotherapy to all sites of disease. For lesions less than 4.5 cm, traditional SBRT will be used. For sites 4.5 cm or greater, Lattice SBRT will be used. For Lattice SBRT, radiotherapy will be prescribed to 20 Gy in 5 fractions delivered every other day with a LATTICE simultaneous integrated boost (SIB) to 66.7 Gy in 5 fractions.
  Interventions: Radiation: Lattice stereotactic body radiation therapy

INTERVENTIONS:
Radiation: Lattice stereotactic body radiation therapy — For Lattice SBRT, the daily prescription dose will be 20 Gy to be delivered to the PTV_2000 with a simultaneous integrated boost of 66.7 Gy to be delivered to the PTV_6670 over 5 fractions (4 Gy and 13.2 Gy to the PTV_2000 and PTV_6670, respectively).
  Other Names: Lattice SBRT

SUMMARY:
Unresectable (including metastatic) conventional chondrosarcoma requires high dose radiation for local control. Radiation Oncologists have traditionally used long radiation courses and concern for toxicity to surrounding organs at risk. Stereotactic body radiation therapy (SBRT) has the ability to deliver high doses of radiation in a manner that may improve clinical response but has size limitations. SBRT delivered with lattice radiotherapy (LRT) may safely dose escalate smaller portions of the tumor and also provide improved cancer control. This study is to evaluate the safety and initial efficacy of this treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed conventional chondrosarcoma.
* At least one, large targetable lesion defined as: 1 lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 45 mm with radiographic imaging or with calipers by clinical exam.
* Deemed metastatic and/or unresectable by multidisciplinary review. Patients with prior resection with gross residual disease that are subsequently deemed ineligible for further resection are allowed.
* Patients that have had prior chemotherapy are allowed
* At least 14 years of age
* ECOG performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
* Radiotherapy is known to be teratogenic. For this reason women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 6 months after completion of the study
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Dedifferentiated chondrosarcoma and extra-skeletal myxoid chondrosarcoma are excluded.
* Patients with greater than 5 measurable metastatic lesions as determined by multidisciplinary review are excluded
* Prior radiotherapy that overlaps with any planned site of protocol radiotherapy.
* Currently receiving any systemic cancer therapy agents. Systemic therapy prior to radiotherapy or planned after radiotherapy delivery are allowed at the discretion of the treating radiation oncologist.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 20 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended. Recommend exclusion of specific ART agents based on predicted drug-drug interactions (i.e. for sensitive CYP3A4 substrates, concurrent strong CYP3A4 inhibitors (ritonavir and cobicistat) or inducers (efavirenz) should be contraindicated).

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related grade 3 or higher non-hematologic adverse events | From start of treatment through 90 days post-treatment (approximately 3.5 months)
  -As scored by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Spraker, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu